CLINICAL TRIAL: NCT03198676
Title: A Single Centre, Partially Blinded, Randomised Study to Compare the Effect of Two PrEP-001 Nasal Powder Formulations on Nasal Mucosa and Serum Cytokine Production in Healthy Human Volunteers
Brief Title: A Safety Study to Compare the Effect of Two PrEP-001 Nasal Powder Formulations on Nasal Mucosa and Serum Cytokine Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prep Biopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: PrEP-001-104
Record Dates: First submitted 2017-06-15; First posted 2017-06-26 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Poly I-C

STUDY DESIGN:
Intervention Model Description: Randomised partially blinded, partially placebo controlled, repeat dose
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A - PrEP-001 6.4 mg - 0.8 mg/spray (Active Comparator): PrEP-001 Nasal Powder, 0.8 mg/spray (G-006) (Formulation A)
  Interventions: Drug: PrEP-001 6.4 mg
- B - PrEP-001 6.4 mg - 1.6 mg/spray (Active Comparator): PrEP-001 Nasal Powder, 1.6 mg/spray (F002) (Formulation B)
  Interventions: Drug: PrEP-001 6.4 mg
- C - PrEP-001 3.2 mg - 1.6 mg/spray (Active Comparator): PrEP-001 Nasal Powder, 1.6 mg/spray (F002) (Formulation B)
  Interventions: Drug: PrEP-001 3.2 mg
- D - Placebo (Placebo Comparator): PrEP-001 Placebo Nasal Powder (matching Formulation B)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PrEP-001 6.4 mg — 6.4 mg as 4 sprays per nostril (ie total of 8 sprays for a single dose) using Aptar unit dose strength powder (UDSP) device
  Other Names: Poly-IC
  Arms: A - PrEP-001 6.4 mg - 0.8 mg/spray
Drug: PrEP-001 6.4 mg — 6.4 mg as 2 sprays per nostril (ie total of 4 sprays for a single dose) using Aptar UDSP device
  Other Names: Poly-IC
  Arms: B - PrEP-001 6.4 mg - 1.6 mg/spray
Drug: PrEP-001 3.2 mg — 3.2 mg as 1 spray per nostril (ie total of 2 sprays for a single dose) using Aptar UDSP device
  Other Names: Poly-IC
  Arms: C - PrEP-001 3.2 mg - 1.6 mg/spray
Drug: Placebo — 2 sprays per nostril (ie total of 4 sprays for a single dose) using Aptar UDSP device
  Arms: D - Placebo

SUMMARY:
A safety study to compare the effect of two different formulations of PrEP-001 nasal powder when dosed in healthy subjects

DETAILED DESCRIPTION:
A single centre, randomised, partially blinded placebo-controlled repeat dose study in healthy male subjects to compare the effect of two different formulations of PrEP-001 nasal powder on nasal mucosal and serum cytokine profiles when dosed for up to five days in health subjects and provide additional safety and tolerability information on active PrEP-001 nasal powder.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged 18 to 65 years
* A body weight of >50 kg and body mass index .18.0 to <32.0 kg/m2
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months. A confirmed positive urine cotinine test at screening and admission
* Current smokers of e-cigarettes and nicotine replacement products and those who have smoked these products within the last 12 months
* Subject who have significant history of any tobacco use at any time (total ≥10 pack years history)
* Subjects who do not have suitable veins for multiple venepunctures as assessed by the investigator at screening
* Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1)
* Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1)
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder, as judged by the investigator
* Any chronic medical condition that could significantly reduce the ability of the subject to participate in the study or pose a safety concern eg unstable angina, uncontrolled diabetes mellitus, anaemia
* Any concurrent serious illness (eg diagnosis of severe depression, pulmonary hypertension, history of malignancy) that may interfere with a subject completing the study. Basal cell carcinoma within 5 years of initial diagnosis or with evidence of recurrence is also an exclusion
* Any finding in the medical history review, physical examination (including nasal exam with nasal speculae), screening investigations, that in the opinion of the investigator would compromise the subject's ability to safely complete the study
* Has experienced upper or lower respiratory infection (viral, fungal or bacterial) that resolved less than 4 weeks before Day 1
* Has required antibiotic treatment for a lower respiratory tract infection in the 3 months prior to the study
* Subjects with a significant nasal condition eg Wegener's granulomatosis, that could interfere with study assessments
* Any significant abnormality altering the anatomy of the nose or nasopharynx on examination
* Any nasal or sinus surgery within 6 months of Day 1
* Any clinically significant history of epistaxis (nosebleeds) within the last 12 months and/or history of being hospitalised due to epistaxis on any previous occasion
* History or evidence of autoimmune disease or known immunodeficiency of any cause - with the exception of atopic eczema/atopic dermatitis. Subjects with clinically mild atopic eczema/atopic dermatitis may be included at the Investigator's discretion (eg if there is no regular use of topical steroids, no eczema in cubital fossa)
* Subjects with known history of Immunosuppression or known chronic viral infection
* Has active seasonal or perennial nasal/pharyngeal allergies at screening visit; or anticipates to have such symptoms during the study duration; or has had symptoms in the 4 weeks prior to Day 1
* Presence or history of clinically significant allergy requiring treatment (including food or drug allergy), as judged by the investigator
* Known allergy or adverse reaction history to formulation components
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration (see Section 11.4). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Changes in baseline in nasal mucosal secretions and serum cytokine concentrations | 5 days
  Changes from baseline in nasal mucosal secretions and serum cytokine concentrations when dosed for up to 5 days with 2 different formulations of PrEP 001 Nasal Powder (ie 6.4 mg Formulation B vs 6.4 mg Formulation A)

SECONDARY OUTCOMES:
Changes in baseline in nasal mucosal secretions and serum cytokine concentrations | 5 days
  Changes from baseline in nasal mucosal secretions and serum cytokine concentrations when dosed for up to 5 days with PrEP 001 Nasal Powder 6.4 mg Formulation B and matching placebo Formulation B
Changes in baseline in nasal mucosal secretions and serum cytokine concentrations | 5 days
  Changes from baseline in nasal mucosal secretions and serum cytokine concentrations when dosed for up to 5 days with PrEP-001 Nasal Powder (3.2 mg and 6.4 mg Formulation B
Assessment of safety parameters | 5 days
  Assessment of the following safety variables: physical examination, safety laboratory tests, vital signs, ECGs and AEs (Formulation B vs Formulation A)

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MBChB BSc, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No